Official Title: A Randomized, Double-Blind, Vehicle-Controlled Study of the Efficacy and Safety of

Ruxolitinib Cream in Participants With Cutaneous Lichen Planus

NCT Number: NCT05593432

**Document Date:** Statistical Analysis Plan: 30-Aug-2023

# **Statistical Analysis Plan**



## INCB 18424-216

A Phase 2, Randomized, Double-Blind, Vehicle-Controlled, Study of the Efficacy and Safety of Ruxolitinib Cream in Participants With Cutaneous Lichen Planus

| IND Number: | 77,101 |
|---|---|
| Sponsor: | Incyte Corporation 1801 Augustine Cut-Off Wilmington, DE 19803 United States |
| <b>Protocol Version:</b> | Protocol Amendment 1 dated 27 MAR 2023 |
| <b>CRF Approval Date:</b> | 20 JUL 2023 |
| SAP Version: | Original |
| SAP Author: | PhD |
| Date of Plan: | 30 AUG 2023 |

This study is being conducted in compliance with Good Clinical Practice, including the archiving of essential documents.

# **TABLE OF CONTENTS**

| TITLE I | PAGE | 1 |
|---------|-------------------------------------------------------------|----|
| TABLE | OF CONTENTS | 2 |
| LIST O | F ABBREVIATIONS | 6 |
| 1. | INTRODUCTION | 8 |
| 2. | STUDY INFORMATION, OBJECTIVES, AND ENDPOINTS | 9 |
| 2.1. | Protocol and Case Report Form Version | 9 |
| 2.2. | Study Objectives and Endpoints | 9 |
| 3. | STUDY DESIGN | 12 |
| 3.1. | Randomization | 12 |
| 3.2. | Control of Type I Error | 12 |
| 3.3. | Sample Size Considerations | 13 |
| 3.4. | Schedule of Assessments | 13 |
| 4. | DATA HANDLING DEFINITIONS AND CONVENTIONS | 14 |
| 4.1. | Scheduled Study Evaluations and Study Periods | 14 |
| 4.1.1. | Day 1 | 14 |
| 4.1.2. | Study Day | 14 |
| 4.1.3. | Baseline Value | 14 |
| 4.1.4. | Handling of Missing and Incomplete Dates | 15 |
| 4.2. | Variable Definitions | 15 |
| 4.2.1. | Body Mass Index | 15 |
| 4.2.2. | Prior and Concomitant Medication | 15 |
| 5. | STATISTICAL METHODOLOGY | 16 |
| 5.1. | General Methodology | 16 |
| 5.2. | Treatment Groups | 16 |
| 5.3. | Analysis Populations | 16 |
| 5.3.1. | Intent-to-Treat Population | 16 |
| 5.3.2. | Safety Population | 16 |
| 5.3.3. | Open-Label Extension Evaluable Population | 16 |
| | | 17 |
| 6. | BASELINE, EXPOSURE, AND DISPOSITION | 17 |
| 6.1. | Demographics, Baseline Characteristics, and Disease History | 17 |

| 6.1.1. | Demographics and Baseline Characteristics | 17 |
|----------|------------------------------------------------------|----|
| 6.1.2. | Baseline Disease Characteristics and Disease History | 17 |
| 6.1.3. | Disease History | 18 |
| 6.1.4. | Medical History | 18 |
| 6.2. | Disposition of Participant | 18 |
| 6.3. | Protocol Deviations | 18 |
| 6.4. | Exposure | 18 |
| 6.5. | Study Drug Compliance | 19 |
| 6.6. | Prior and Concomitant Medication | 19 |
| 7. | EFFICACY | 20 |
| 7.1. | Efficacy Hypotheses | 20 |
| 7.2. | Efficacy Measures | 20 |
| 7.2.1. | Investigator's Global Assessment | 20 |
| | | 21 |
| | | 21 |
| | | 22 |
| 7.2.5. | Body Surface Area | 22 |
| 7.2.6. | Patient-Reported Outcomes | 23 |
| 7.2.6.1. | Itch Numerical Rating Scale | 23 |
| 7.2.6.2. | Skin Pain Numerical Rating Scale | 23 |
| | | 24 |
| | | 24 |
| | | 25 |
| | | 25 |
| | | 25 |
| 7.3. | Analysis of the Primary Efficacy Parameter | 26 |
| 7.3.1. | Primary Efficacy Analysis | 26 |
| 7.3.2. | Subgroup Analyses for Primary Endpoint | 26 |
| 7.4. | Analysis of the Secondary Efficacy Parameters | 26 |
| 7.4.1. | Continuous Efficacy Endpoints | 26 |
| 7.4.2. | Categorical Efficacy Endpoints | 26 |
| 7.4.3. | Time-To-Event Efficacy Endpoint | 27 |

| | | 27 |
|----|------------------------------------------------|----|
| | | 29 |
| | | 29 |
| | | 29 |
| | SAFETY AND TOLERABILITY | 30 |
| | General Considerations | 30 |
| | Adverse Events | 30 |
| | Adverse Event Definitions | 30 |
| | Adverse Event Summaries | 31 |
| | Clinical Laboratory Tests | 32 |
| | Laboratory Value Definitions | 32 |
| | Laboratory Value Summaries | 32 |
| | Vital Signs | 33 |
| | PLANNED ANALYSES | 33 |
| | CHANGES AND MODIFICATIONS TO THE ANALYSIS PLAN | 34 |
| | Changes to Protocol-Defined Analyses | 34 |
| | Changes to the Statistical Analysis Plan | 34 |
| | REFERENCES | 35 |
| 1D | OIX A. PLANNED TABLES, FIGURES, AND LISTINGS | 36 |

## LIST OF TABLES

| Table 1: | Objectives and Endpoints | 9 |
|-----------|----------------------------------------------------------|----|
| | | 20 |
| | | 22 |
| Table 4: | Criteria for Clinically Notable Vital Sign Abnormalities | 33 |
| Table 5: | Statistical Analysis Plan Versions | 34 |
| | LIST OF FIGURES | |
| Figure 1: | Study Design Schema | 12 |

# LIST OF ABBREVIATIONS

| Abbreviation | Term |
|---|---|
| AE | adverse event |
| AIF | area involvement factor |
| ASR | application site reaction |
| BID | twice daily |
| BSA | body surface area |
| CI | confidence interval |
| CRF | case report form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DBVC | double-blind, vehicle-controlled |
| DBVC | double-offind, venicle-controlled |
| eCRF | electronic case report form |
| | erythematous papules |
| Ер | hyperpigmented hypertrophic papules and plaques |
| Hp<br>IGA | Investigator's Global Assessment |
| IGA-TS | Investigator's Global Assessment-Treatment Success (IGA score of 0 or 1 with ≥ 2-grade improvement from baseline) |
| ITCH4 | ≥ 4-Point improvement in Itch NRS score |
| ITT | intent-to-treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MF | multiplication factor |
| NCI | National Cancer Institute |
| NRS | numeric rating scale |
| OLE | open-label extension |
| PIH | postinflammatory hyperpigmentation |
| PT | preferred term |
| rux | ruxolitinib |

| Abbreviation | Term |
|--------------|----------------------------------|
| SAP | Statistical Analysis Plan |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| VC | vehicle-controlled |
| Vp | violaceous flat papules |
| Vpl | violaceous flat plaques |
| WHO | World Health Organization |

#### 1. INTRODUCTION

INCB 18424-216 is a Phase 2, randomized, DBVC study to evaluate the efficacy and safety of ruxolitinib 1.5% cream BID in participants with cutaneous LP over a 16-week treatment period followed by a 16-week OLE period. A 30-day post-treatment safety follow-up visit will be conducted after the OLE period.

The purpose of this SAP is to provide details of the statistical analyses that have been outlined in the INCB 18424-216 Protocol.

## 2. STUDY INFORMATION, OBJECTIVES, AND ENDPOINTS

## 2.1. Protocol and Case Report Form Version

This SAP is based on INCB 18424-216 Protocol Amendment 1 dated 27 MAR 2023 and CRFs approved 20 JUL 2023. Unless superseded by an amendment, this SAP will be effective for all subsequent Protocol amendments and eCRF versions.

## 2.2. Study Objectives and Endpoints

Table 1 presents the objectives and endpoints.

**Table 1:** Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To establish the efficacy of ruxolitinib 1.5% cream BID in participants with cutaneous LP. | • IGA-TS response is defined as an IGA score of 0 or 1 with ≥ 2-grade improvement from baseline at Week 16; this is the proportion of participants achieving IGA-TS at Week 16. |
| Secondary | |
| To further access the treatment effects of ruxolitinib 1.5% cream BID in participants with cutaneous LP. | IGA-TS response at each scheduled postbaseline visit up to and including Week 32 will be the proportion of participants achieving IGA-TS at each scheduled postbaseline visit. |
| | <ul> <li>ITCH4 response is defined as a ≥ 4-point<br/>improvement in Itch NRS score from baseline at<br/>each scheduled postbaseline visit, up to and<br/>including Week 32; it is the proportion of<br/>participants with ITCH4 at each scheduled<br/>postbaseline visit.</li> </ul> |
| | Time to achieve ITCH4. |
| | Change from baseline in the Skin Pain NRS score<br>at each scheduled postbaseline visit, up to and<br>including Week 32. |
| To evaluate the safety and tolerability of ruxolitinib 1.5% cream BID. | The type, frequency, and severity of AEs, including changes in vital signs and clinical laboratory blood samples. |

**Table 1:** Objectives and Endpoints (Continued)

| Objectives | Endpoints |
|------------|-----------|

**Table 1:** Objectives and Endpoints (Continued)



#### 3. STUDY DESIGN

This is a Phase 2, randomized, DBVC study in participants aged  $\geq 18$  years who have predominantly cutaneous LP (covering  $\leq 20\%$  BSA) and baseline IGA score  $\geq 3$ . The study will consist of a 16-week DBVC period followed by a 16-week OLE period.

Approximately 60 participants will be randomized 1:1 to either ruxolitinib 1.5% cream BID or vehicle cream BID. Participants will be stratified by baseline IGA score (3 or 4). Participants will apply either ruxolitinib 1.5% cream BID or vehicle cream BID through Week 16 to all affected areas identified at baseline.

At Week 16, participants who meet the criteria (compliant with the Protocol and without safety concerns) will enter the 16-week OLE period. Participants randomized initially to vehicle cream in the DBVC period will be crossed over to ruxolitinib 1.5% cream BID and participants randomized to ruxolitinib 1.5% cream at baseline will continue to apply ruxolitinib 1.5% cream BID through Week 32. In the OLE period, participants will only treat active lesions up to 20% BSA. At Week 16, the LP treatment area will be evaluated by the investigator to assess the disease and confirm whether treatment continuation is required (IGA score  $\geq$  1) during the OLE period or can otherwise (re)enter an observation/no treatment cycle (IGA score = 0).

The study schema is shown below in Figure 1.

Figure 1: Study Design Schema



The primary analysis will occur after the primary database lock, when all participants have completed the DBVC period. The final analysis will occur when all participants have completed or withdrawn from the study.

#### 3.1. Randomization

Approximately 60 participants will be randomized 1:1 to either ruxolitinib 1.5% cream BID or vehicle cream BID, stratified by baseline IGA score (3 or 4).

## 3.2. Control of Type I Error

The significance level for primary efficacy analysis will be 0.05 for a 2-sided test.

### 3.3. Sample Size Considerations

Approximately 60 participants will be randomized 1:1 (ie, ruxolitinib 1.5% cream BID or vehicle cream BID) and stratified by baseline IGA (3 or 4). The sample size calculation is based on the Fisher exact test for the statistical comparison on the primary efficacy endpoint: the proportion of participants achieving IGA-TS at Week 16. Based on previous studies (INCB 18424-303 and -304) and the results from an investigator sponsored trial (Mangold et al 2021) with topical ruxolitinib (NCT03697460), the preliminary assumption of response rates is 58% for ruxolitinib 1.5% cream and 20% for vehicle cream. Using a 2-sided alpha of 0.05, the sample size, based on the current setup, will have > 80% power to detect a difference between active treatment and vehicle. In addition to providing adequate power for efficacy variables, the sample size is determined to provide an adequate database for safety evaluations.

#### 3.4. Schedule of Assessments

Refer to Protocol Amendment 1 dated 27 MAR 2023 for a full description of all study procedures and assessment schedules for this study.

#### 4. DATA HANDLING DEFINITIONS AND CONVENTIONS

### 4.1. Scheduled Study Evaluations and Study Periods

#### 4.1.1. Day 1

Day 1 is the date that the first application of ruxolitinib cream or vehicle cream in the specific period.

For randomized participants not treated with any study drug, Day 1 is defined as the date of randomization.

### **4.1.2. Study Day**

If a visit/reporting date is on or after Day 1, then the study day at the visit/reporting date will be calculated as

```
Day \# = (visit/reporting date - Day 1 date + 1).
```

If the visit/reporting date is before Day 1, then the study day at the visit/reporting date will be calculated as

```
Day \# = (visit/reporting date - Day 1 date).
```

A study day of -1 indicates 1 day before Day 1.

#### 4.1.3. Baseline Value

Baseline is the last nonmissing measurement obtained before or on the day of the first application of ruxolitinib cream or vehicle cream for the DBVC period.

For randomized participants not treated with any study drug, baseline is defined as the last nonmissing assessment before randomization for all parameters.

For participants who continue in the OLE period, baseline is defined as follows:

- For efficacy evaluation in the OLE period, baseline is the last nonmissing measurement obtained before or on the day of first application of study treatment in the DBVC period.
- For safety evaluation in the OLE period:
  - For participants who cross over from vehicle group to ruxolitinib cream, the
    baseline is the last nonmissing measurement obtained before or on the day of first
    application of ruxolitinib cream in the OLE period.
  - For participants who apply ruxolitinib cream in both periods, baseline is the last nonmissing measurement obtained before or on the day of first application of study treatment in the DBVC period.

When a scheduled assessment and an unscheduled assessment occur on the same day and the times of the assessments are not available, use the following convention to determine baseline:

- If both a scheduled and an unscheduled visit are available on the day of the first dose and the time is missing, use the scheduled assessment as baseline.
- If all scheduled assessments are missing on the day of the first application, but an unscheduled assessment is available, use the unscheduled assessment as baseline.

### 4.1.4. Handling of Missing and Incomplete Dates

In general, values for missing dates will not be handled unless methods for handling missing dates are specified in this section or relevant sections. The original reported dates collected on the eCRF should be used in all relevant listings. The following rules will be used for handling partial dates for analyses requiring dates.

Partial LP diagnosis date will be handled as follows:

- If only the day is missing, then the fifteenth of the month will be used.
- If both the month and day are missing, then 01 JUL of the year will be used.
- If the diagnosis date is completely missing, then the time since diagnosis will not be calculated.

#### 4.2. Variable Definitions

### 4.2.1. Body Mass Index

Body mass index will be calculated as follows:

Body mass index  $(kg/m^2) = [weight (kg)] / [height (m)]^2$ 

#### 4.2.2. Prior and Concomitant Medication

Prior medication is defined as any nonstudy medication started before the first application of ruxolitinib 1.5% cream BID or vehicle cream BID.

Concomitant medication is defined as any nonstudy medication that is started accordingly:

- Before the date of first application of ruxolitinib 1.5% cream or vehicle cream and is ongoing throughout the study or ends on/after the date of first study drug application.
- On/after the date of first application of ruxolitinib 1.5% cream or vehicle cream and is ongoing or ends during the course of study.

A prior medication could also be classified as "both prior and concomitant medication" if the end date is on or after first application of ruxolitinib 1.5% cream or vehicle cream. In the listing, it will be indicated whether a medication is only prior, only concomitant, or both prior and concomitant.

For the purposes of analysis, all medications will be considered concomitant medications unless the medications can unequivocally be defined as not concomitant.

#### 5. STATISTICAL METHODOLOGY

### **5.1.** General Methodology

Unless otherwise noted, SAS® software (SAS Institute Inc, Cary, NC; v9.4 or later) will be used for the generation of all tables, graphs, and statistical analyses. Descriptive summaries for continuous variables will include, but not be limited to, the number of observations, mean, standard deviation, median, minimum, and maximum. Descriptive summaries for categorical variables will include the number and percentage of participants in each category.

### **5.2.** Treatment Groups

This is a randomized, DBVC study followed by an OLE period. Table summaries, unless otherwise indicated, will present data by treatment group.

For the DBVC period, the treatment groups will be vehicle cream and ruxolitinib 1.5% cream.

For the OLE period, the participants will be grouped according to the treatment they received during the DBVC period:

- Vehicle cream to ruxolitinib 1.5% cream
- Ruxolitinib 1.5% cream

## 5.3. Analysis Populations

### **5.3.1.** Intent-to-Treat Population

All participants who are randomized will constitute the ITT population. Treatment groups for this population will be defined according to the treatment assignment at the time of randomization regardless of the actual study drug the participant might take during their participation in the DBVC period.

The ITT population will be used for the summary of demographics, baseline characteristics, participant disposition, and analyses of all efficacy data.

### **5.3.2.** Safety Population

The safety population will include all participants who applied ruxolitinib 1.5% cream BID or vehicle cream BID at least once. Treatment groups for this population will be determined according to the actual treatment the participant applied on Day 1 regardless of assigned study drug treatment.

All safety analyses will be conducted using the safety population.

### **5.3.3.** Open-Label Extension Evaluable Population

All analyses for the OLE period will be conducted with the OLE evaluable population, which includes all participants who applied ruxolitinib 1.5% cream at least once during the OLE period.

### 6. BASELINE, EXPOSURE, AND DISPOSITION

Appendix A provides a list of planned tables, figures, and listings. Sample data displays are included in a separate document.

### 6.1. Demographics, Baseline Characteristics, and Disease History

#### 6.1.1. Demographics and Baseline Characteristics

The following demographics and baseline characteristics will be summarized by treatment groups and overall for the ITT population in the DBVC period and for the OLE evaluable population in the OLE period: age, sex, race, ethnicity, weight, height, and body mass index.

### 6.1.2. Baseline Disease Characteristics and Disease History

For the ITT population, the baseline disease characteristics will be summarized by treatment group and will include, but not limited to, the following:

- Disease duration (years)
- LP diagnosis confirmed by previous biopsy (yes/no)
- Anatomic location (hands/wrists, forearms/arms, neck, face, ankle/feet, legs, back/buttocks, chest, abdomen, mucosal-mouth, mucosal-nose, mucosal-vulva/vagina, mucosal-esophagus, or other)
- Variant (type) of LP (hypertrophic LP, annular LP, bullous LP, actinic LP, LP pigmentosus, inverse LP, atrophic LP, lichen planopilaris [follicular LP], nail LP, mucosal LP-oral, mucosal LP-genital, mucosal LP-esophageal, mucosal LP-otic, indeterminate/unspecified, unknown, or other)
- Family history of LP (yes/no)
- History of skin infection related to LP requiring antibiotic treatment (yes/no)
- History of other skin diseases (yes/no)
- Days since onset of current episode of LP flare/activity
- Number of flares/episodes of LP in the past year other than current flare the participant experienced
- Clinical manifestations related to LP (% participants with each of the manifestations)
- Prior treatment received for LP (yes/no)

- Skin type using Fitzpatrick classification (Type I through VI)
- Total % BSA affected
- Baseline IGA score
- Baseline Itch NRS score
- Baseline Skin Pain NRS

### **6.1.3.** Disease History

The time since disease duration will be summarized for all participants in the ITT population.

Time since diagnose (ie, disease duration [years]) will be calculated as follows:

Disease duration (years) = (date of randomization – date of initial LP diagnosis +1) / 365.25.

#### 6.1.4. Medical History

For participants in the ITT population during the DBVC period, medical history will be summarized by assigned treatment groups. This summary will include the number and percentage of participants with medical history for each body system/organ class as documented on the eCRF.

### 6.2. Disposition of Participant

The number and percentage of participants who were randomized, treated, and completed the DBVC period, as well as the number and percentage of participants who discontinued the treatment or withdrew from the study during the DBVC period with a primary reason for discontinuation, will be summarized as part of the ITT population.

The number and percentage of participants who completed the OLE period, in addition to those participants who discontinued treatment or withdrew from the study during the OLE period with a primary reason for discontinuation, will be summarized as part of the OLE evaluable population.

#### 6.3. Protocol Deviations

Protocol deviations will be summarized and listed by treatment group and overall for ITT and OLE populations.

### 6.4. Exposure

For participants in the safety population in the DBVC period, the OLE evaluable population in the OLE period, and those who applied ruxolitinib 1.5% cream BID throughout the study, study drug exposure will be summarized by treatment group, descriptively, as follows:

• Duration of treatment (days):

Date of last application of ruxolitinib cream or vehicle cream in the specific period – date of first application of ruxolitinib cream or vehicle cream in the specific period + 1

• Total amount of cream applied (g):

Total weight of ruxolitinib cream or vehicle cream dispensed in the specific period – total weight of ruxolitinib cream or vehicle cream returned in the specific period

• Average daily application:

Total amount of cream applied in the specific period (g) / [duration of treatment with study cream in the specific period (days) – number of interrupted days with study cream in the specific period].

## 6.5. Study Drug Compliance

The overall compliance (%) for the application of ruxolitinib 1.5% cream BID or vehicle cream BID during the DBVC period will be calculated for all participants in the safety population as follows:

Cream application compliance (%) =  $100 \times [\text{total number of nonmissing applications}] / [\text{total number of intended applications}], where$ 

Total number of nonmissing applications = number of applications that the participants actually applied during the study, and

Total number of intended applications =  $2 \times \text{duration of treatment (days)} - \text{number of interrupted applications.}$ 

#### 6.6. Prior and Concomitant Medication

Prior medications and concomitant medications will be coded using the WHO Drug Dictionary. The number and percentage of participants with prior and concomitant medication will be summarized by treatment group, as well as overall for the ITT population during the DBVC period by WHO drug class and WHO drug preferred term. For the OLE period, only concomitant medications will be summarized based on OLE evaluable population.

#### 7. EFFICACY

Appendix A provides a list of data displays. Sample data displays are included in a separate document.

### 7.1. Efficacy Hypotheses

The primary hypothesis is the superiority of ruxolitinib 1.5% cream BID compared with vehicle cream BID in the proportion of participants achieving IGA-TS at Week 16.

## 7.2. Efficacy Measures

### 7.2.1. Investigator's Global Assessment

The IGA to assess cutaneous LP has been modified by the sponsor to appropriately assess LP. The investigator/rater will assess the lesions at the study visits by using the descriptors that best describe the overall appearance of the lesions at a given timepoint. It is not necessary that all characteristics under the morphological description be present.

The IGA-TS is defined as an IGA score of 0 or 1 with  $\geq$  2-grade improvement from baseline. Nonresponder imputation will be used to handle missing postbaseline values in the DBVC period.





### 7.2.5. Body Surface Area

The total % BSA affected will be estimated at each visit. The BSA assessment will be approximated to the nearest 0.1% using the Palmar Method as a guide, which is the palm plus 5 digits, with fingers tucked together and thumb tucked to the side (handprint) as 1% BSA and the thumb as 0.1% BSA.

#### 7.2.6. Patient-Reported Outcomes

Patient-reported outcomes will be collected and assessed. For all patient-reported outcome assessments conducted at the study site, in order to avoid bias in the participants' responses to the questionnaires, assessments will be completed before any other evaluations or study procedures on the day of the study visit and prior to any treatment-related discussions with the investigator or study site staff.

#### 7.2.6.1. Itch Numerical Rating Scale

The Itch NRS is a daily participant-reported measure (24-hour recall) of the worst level of itch intensity (Kimball et al 2016, Silverberg et al 2021). Participants will be instructed to complete and record their Itch NRS in a diary each evening beginning on the day of screening through Week 32 or treatment discontinuation, whichever comes first. Participants will rate itch severity of their LP by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best describes the worst level of itch they experienced in the past 24 hours.

The participant's baseline Itch NRS score will be determined by averaging the 7 daily NRS scores before Day 1 (ie, Days –7 to –1) for all the by-visit summaries. The by-visit Itch NRS score for postbaseline visits will be determined by averaging the 7 daily NRS scores before the visit day. If 4 or more daily scores (out of the 7) are missing, the by-visit Itch NRS score will be set to missing. For all daily itch-related analyses, including time to achieve Itch NRS score improvement of at least 4 points analysis, baseline will be defined as the last available Itch NRS score during the week prior to Day 1 (ie, Days –7 to –1). Nonresponder imputation will be used to handle missing postbaseline values in the DBVC period.

A participant is said to have an ITCH4 response if they achieved a  $\geq$  4-point improvement in Itch NRS score from baseline. For determining ITCH4 response at a visit, the by-visit Itch NRS score will be compared with the baseline Itch NRS score. For the endpoint time to achieve ITCH4, the daily Itch NRS score will be compared with the baseline Itch NRS score.

#### 7.2.6.2. Skin Pain Numerical Rating Scale

Participants will be instructed to complete and record the Skin Pain NRS in a diary each evening beginning on the day of screening through Week 32 or treatment discontinuation. Participants will rate their pain, which will include all types of pain (eg, burning, tearing, pulling, stabbing, etc) severity of the LP by selecting a number from 0 (no pain) to 10 (worst imaginable pain) that best describes the worst level of pain they experienced in the past 24 hours.

The participant's baseline Skin Pain NRS score will be determined by averaging the 7 daily NRS scores before Day 1 (ie, Days –7 to –1). The by-visit Skin Pain NRS score for postbaseline visits will be determined by averaging the 7 daily NRS scores before the visit day. If 4 or more daily scores (out of the 7) are missing, the Skin Pain NRS score at the visit will be set to missing. No imputation will be performed for missing values.





### 7.3. Analysis of the Primary Efficacy Parameter

### 7.3.1. Primary Efficacy Analysis

The primary efficacy analysis will be based on the ITT population. The primary efficacy endpoint is the IGA-TS response, defined as an IGA score of 0 or 1 with  $\geq$  2-grade improvement from baseline, at Week 16. The comparison of the proportions of participants achieving IGA-TS at Week 16 will be made between the ruxolitinib 1.5% cream BID arm and the vehicle cream BID arm. The primary hypothesis (the superiority of ruxolitinib 1.5% cream BID compared with vehicle cream BID in participants with cutaneous LP) will be tested using a Cochran-Mantel-Haenszel test stratified by baseline IGA score (3 or 4) at a 2-sided  $\alpha = 0.05$  level. The p-value and stratum-adjusted IGA-TS response rate difference with 95% CI will be provided. A summary of IGA-TS rates will be reported for each treatment group. Nonresponder imputation will be used to handle missing postbaseline values in the DBVC period.

### 7.3.2. Subgroup Analyses for Primary Endpoint

Subgroups will be formed based on the following participant characteristics and baseline variables for those participants whose data are available:

- Sex: female versus male
- Baseline categorical age:  $\geq 18$  and < 65 versus  $\geq 65$
- Baseline duration of disease:  $\leq 1, > 1$  and  $\leq 5, > 5$
- Race: Black/African American versus White/Asian/other

The primary efficacy endpoint will be summarized using descriptive statistics based on the ITT population for the aforementioned subgroups.

## 7.4. Analysis of the Secondary Efficacy Parameters

All secondary efficacy analyses will be conducted for the ITT population.

#### 7.4.1. Continuous Efficacy Endpoints

Summary statistics for the following continuous measurements, including change from baseline, will be presented for each treatment arm:

• By-visit Skin Pain NRS score

The summary statistics, including sample size, mean, median, standard deviation, minimum, maximum, first quartile, third quartile, and 95% CI, will be presented by visit.

### 7.4.2. Categorical Efficacy Endpoints

For the following categorical parameters, summary statistics, including sample size, frequency, and percentages, will be presented by visit.

- IGA-TS response
- By-visit ITCH4 response

In addition, a Cochran-Mantel-Haenszel test stratified by baseline IGA score (3 or 4) at a 2-sided  $\alpha = 0.05$  level will be used for the comparison between ruxolitinib 1.5% cream BID and vehicle cream BID at Week 16 for ITCH4 response. The p-value and stratum-adjusted response rate difference with 95% CI will be provided.

#### 7.4.3. Time-To-Event Efficacy Endpoint

The time to achieve Itch NRS score improvement of at least 4 points from baseline (ie, ITCH4) will use the daily Itch NRS score in comparison to baseline Itch NRS score in the DBVC period. A log-rank test stratified by randomization stratification factor, baseline IGA score (3 or 4), will be used for between-treatment group comparisons. The hazard ratio and its 95% CI will be estimated based on the stratified Cox regression model using Efron's method accounting for ties. Kaplan-Meier curves will be presented by treatment groups. The number of participants, number of participants with events, and number of participants censored will be summarized by treatment group. The Kaplan-Meier estimate of median time will be presented with its 95% CI. The 95% CI will be calculated using the method by Brookmeyer and Crowley (1982).

The last available value for time to ITCH4 during the DBVC period is the last nonmissing measurement obtained after the first application of study cream and within 30 days after the last application of study cream in DBVC period, or before the first application of study cream in the OLE period, whichever is earlier.







#### 9. SAFETY AND TOLERABILITY

Appendix A provides a list of data displays.

#### 9.1. General Considerations

The analyses in this section will be provided for the safety population in the DBVC period and the OLE evaluable population in the OLE period, unless otherwise specified. Summary tables may be replaced with listings when appropriate. For instance, an AE frequency table may be replaced with a listing if it only contains a few unique preferred terms reported on relatively few participants.

#### 9.2. Adverse Events

#### 9.2.1. Adverse Event Definitions

A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first application of study drug and within 30 days of the last application of study drug. For participants who cross over treatments, the first application date is period-specific; however, the end date is 30 days after the last application date in this period, or the first application date in the next period, whichever comes first. Analysis of AEs (as discussed below) will be limited to TEAEs, but data listings will include all AEs regardless of their timing in relation to study drug application.

Adverse events will be tabulated by MedDRA PT and SOC. Severity of AEs will be graded using the NCI CTCAE v5. The CTCAE reporting guidelines and grading details are available on the Cancer Therapy Evaluation Program website.

The subset of AEs considered by the investigator to be related to study drug will be considered to be treatment-related AEs. If the investigator does not specify the relationship of the AE to study drug, the AE will be considered to be treatment-related. The incidence of AEs and treatment-related AEs will be tabulated. In addition, serious TEAEs will also be tabulated.

Any missing onset date, causality, or severity must be queried for resolution. Unresolved missing causality and severity will be handled according to the following rules:

- An unresolved missing causality will be considered treatment-related.
- An unresolved missing severity will be identified as an unknown severity.

For purposes of analysis, all AEs will be considered TEAEs unless the AE can unequivocally be defined as not treatment-emergent.

Application site reactions are AEs that occur at the site of drug application. A summary of ASRs will be provided.

#### 9.2.2. Adverse Event Summaries

An overall summary of AEs by treatment group will include the following:

- Number (%) of participants reporting any TEAEs
- Number (%) of participants reporting any serious TEAEs
- Number (%) of participants reporting any Grade 3 or higher TEAEs
- Number (%) of participants reporting any treatment-related TEAEs
- Number (%) of participants who temporarily interrupted study treatment because of TEAEs
- Number (%) of participants who permanently discontinued study treatment because of TEAEs
- Number (%) of participants who had any fatal TEAEs

The following summaries will be produced by MedDRA term (if 2 or fewer participants appear in a table, a listing may be appropriate):

- Summary of TEAEs by MedDRA SOC and PT
- Summary of TEAEs by MedDRA PT in decreasing order of frequency
- Summary of TEAEs by MedDRA SOC, PT, and maximum severity
- Summary of TEAEs by MedDRA SOC, PT, and CTCAE grade category
- Summary of Grade 3 or higher TEAEs by MedDRA SOC and PT
- Summary of Grade 3 or higher TEAEs by MedDRA PT in decreasing order of frequency
- Summary of serious TEAEs by MedDRA SOC and PT
- Summary of serious TEAEs by MedDRA PT in decreasing order of frequency
- Summary of treatment-related TEAEs by MedDRA SOC and PT
- Summary of treatment-related TEAEs by MedDRA PT in decreasing order of frequency
- Summary of Grade 3 or higher treatment-related TEAEs by MedDRA SOC and PT
- Summary of treatment-related serious TEAEs by MedDRA SOC and PT
- Summary of TEAEs with a fatal outcome by MedDRA SOC and PT
- Summary of TEAEs leading to dose interruption by MedDRA SOC and PT
- Summary of TEAEs leading to discontinuation of study drug by MedDRA SOC and PT
- Summary of ASR by MedDRA PT in decreasing order of frequency

### 9.3. Clinical Laboratory Tests

### 9.3.1. Laboratory Value Definitions

All laboratory assessments will be performed using a central laboratory with the exception of urine pregnancy tests. Laboratory values and change from baseline values will be summarized descriptively by visit; non-numeric test values will be tabulated when necessary. Baseline will be determined according to Section 4.1.3, using the last nonmissing value collected before the first application, prioritizing scheduled assessments for baseline identification over unscheduled visits. The last record before application in the highest priority will be considered the baseline record. For baseline laboratory candidates with the same date and time in the same priority category, additional rules may be provided after consultation with the medical monitor to delineate which value will be defined as baseline.

### 9.3.2. Laboratory Value Summaries

All test results and associated normal ranges from central laboratories will be reported in SI units. All tests with numeric values will have a unique unit per test. Any laboratory test results and associated normal ranges from local laboratories will be converted to SI units.

When there are multiple laboratory nonmissing values for a participant's particular test at a scheduled visit, central laboratory values have higher priority over local laboratory values. If a tie still exists, the laboratory value with the smallest laboratory sequence number will be used in by-visit summaries.

For test results that will be summarized with available normal ranges, the number and percentage of participants with the laboratory values being low (but never high), normal, high (but never low), and both low and high will be calculated for each test. A shift summary will be produced for each test. The denominator for the percentage calculation will use the number of participants in the baseline category (ie, low, high, normal, or missing) as the denominator for the percentage in each of the categories during the study.

Severity grades will be assigned to laboratory test values based on the numerical component of CTCAE v5. Shift tables will also be presented showing change in CTCAE grade from baseline to the worst grade postbaseline. Separate summaries for abnormally high and abnormally low laboratory values will be provided when the laboratory parameter has both high and low grading criteria. The denominator for the percentage calculation will be the number of participants in the baseline category. The number of participants who experienced worsening of laboratory abnormalities will be summarized by maximum severity.

### 9.4. Vital Signs

Values at each scheduled visit, change, and percentage change from baseline for vital signs, including systolic blood pressure, diastolic blood pressure, pulse, temperature, and respiratory rate will be summarized descriptively.

Normal ranges for vital sign values are defined in Table 4. For participants exhibiting vital sign abnormalities, the abnormal values will be listed along with their assigned treatment group. Alert vital signs are defined as an absolute value outside the defined normal range and percentage change greater than 25%. The abnormal values for participants exhibiting alert vital sign abnormalities will be listed.

**Table 4:** Criteria for Clinically Notable Vital Sign Abnormalities

| Parameter | High Threshold | Low Threshold |
|--------------------------|------------------|-----------------|
| Systolic blood pressure | > 155 mmHg | < 85 mmHg |
| Diastolic blood pressure | > 100 mmHg | < 40 mmHg |
| Pulse | > 100 bpm | < 45 bpm |
| Temperature | > 38°C | < 35.5°C |
| Respiratory rate | > 20 breaths/min | < 8 breaths/min |

#### 10. PLANNED ANALYSES

No formal interim analysis is planned in this study.

There are 2 formal planned analyses:

- The primary analysis will occur after the primary database lock, when all participants have completed the DBVC period. The sponsor will be unblinded after the primary database lock; however, investigators and participants will remain blinded to the individual study treatment assignment after the primary database lock.
- The final analysis will occur when all participants have completed or withdrawn from the study.

# 11. CHANGES AND MODIFICATIONS TO THE ANALYSIS PLAN

All versions of the SAP are listed in Table 5.

**Table 5:** Statistical Analysis Plan Versions

| SAP Version | Date |
|-------------|-------------|
| Original | 30 AUG 2023 |





# 11.2. Changes to the Statistical Analysis Plan

Not applicable.

# 12. REFERENCES

| Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics 1982;38:29-41. |
|---|
| Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther 2004;27:26-35. |
| Kimball AB, Naegeli AN, Edson-Heredia E, et al. Psychometric properties of the Itch Numeric Rating Scale in patients with moderate-to-severe plaque psoriasis. Br J Dermatol 2016;175:157-162. |
| Mangold A, Brumfiel CM, Patel MH, Severson KJ, Zhang N, Pittelkow MR. Ruxolitinib cream in the treatment of cutaneous lichen planus. J Am Acad Dermatol 2021;85(suppl):AB10 [abstract 25713]. |
| Ruxolitinib Cream Investigator's Brochure. Wilmington, DE: Incyte Corporation. |

## APPENDIX A. PLANNED TABLES, FIGURES, AND LISTINGS

This appendix provides a list of the planned tables, figures, and listings for the Clinical Study Report. Shells are provided in a separate document for tables that are not in the most current Standard Safety Tables v1.13.

The lists of tables, figures, and listings are to be used as guidelines. Modifications of the lists that do not otherwise affect the nature of the analysis will not warrant an amendment to the SAP.

#### **Tables**

| Table No. | Title | Population | Standard |
|---|---|---|---|
| Baseline an | nd Demographics Characteristics | | |
| 1.1 Disposi | tion | | |
| 1.1.1 | Analysis Populations | ITT | X |
| 1.1.2.1 | Summary of Participant Disposition in the DBVC Period | ITT | X |
| 1.1.2.2 | Summary of Participant Disposition in the OLE Period | OLE | X |
| 1.1.3 | Summary of Number of Participants Enrolled by Country and Site | ITT | X |
| 1.1.4.1 | Summary of Protocol Deviations in the DBVC Period | ITT | X |
| 1.1.4.2 | Summary of Protocol Deviations in the OLE Period | OLE | X |
| 1.2 Demogr | raphics and Baseline Characteristics | | |
| 1.2.1 | Summary of Demographics and Baseline Characteristics in the DBVC Period | ITT | X |
| 1.2.2 | Summary of Demographics and Baseline Characteristics in the OLE Period | OLE | X |
| 1.3 Baselin | e Disease Characteristics | l | |
| 1.3.1 | Summary of Baseline Disease Characteristics in the DBVC Period | ITT | X |
| 1.3.2 | Summary of Baseline Disease Characteristics in the OLE Period | OLE | X |
| 1.4 Prior a | nd Concomitant Medication | • | |
| 1.4.1 | Summary of Prior Medications in the DBVC Period | ITT | X |
| 1.4.2.1 | Summary of Concomitant Medications in the DBVC Period | ITT | X |
| 1.4.2.2 | Summary of Concomitant Medications in the OLE Period | OLE | X |
| 1.5 Others | 1.5 Others | | |
| 1.5 | Summary of General Medical History in the DBVC Period | ITT | X |
| Efficacy | | | |
| 2.1 IGA Sc | ore | | |
| 2.1.1 | Summary and Analysis of Participants Achieving IGA-TS in Treatment Periods | ITT | |
| 2.1.2 | Summary and Analysis of Participants Achieving IGA-TS by Sex in Treatment Periods | ITT | |
| 2.1.3 | Summary and Analysis of Participants Achieving IGA-TS by Categorical Age in Treatment Periods | ITT | |
| 2.1.4 | Summary and Analysis of Participants Achieving IGA-TS by Duration of Disease in Treatment Periods | ITT | |
| | L | | · |

| Table No. | Title | Population | Standard |
|---|---|---|---|
| 2.1.5 | Summary and Analysis of Participants Achieving IGA-TS by Race in Treatment Periods | ITT | |
| 2.1.6 | Summary of Participants in Each Category of IGA in Treatment Periods | ITT | |
| 2.2 Itch NF | RS Score | | |
| 2.2.1 | Summary of Participants Achieving ITCH4 in Treatment Periods | ITT | |
| 2.2.2 | Summary of By-Visit Itch NRS Score in Treatment Periods | ITT | |
| 2.2.3 | Summary of Daily Itch NRS Score from Day 1 to Day 28 | ITT | |
| 2.2.4 | Summary of Time to ITCH4 in the DBVC Period | ITT | |
| 2.3 Skin Pa | nin NRS Score | - | • |
| 2.3.1 | Summary of By-Visit Skin Pain NRS Score in Treatment Periods | ITT | |
| | | | <u>I</u> |
| | | | T |
| | | | Ι |
| | | | <u> </u> |
| - 10 = - · | | | |
| 2.13 BSA | T | | <u> </u> |
| 2.13.1 | Summary of Total % BSA in Treatment Periods | ITT | |
| Safety | | | |
| _ | re & Compliance | | T |
| 3.1.1.1 | Summary of Exposure in the DBVC Period | Safety | X |
| 3.1.1.2 | Summary of Exposure in the OLE Period | OLE | X |

| Table No. | Title | Population | Standard |
|---|---|---|---|
| 3.1.1.3 | Summary of Exposure in Treatment Periods | Safety | X |
| 3.1.2.1 | Summary of Study Drug Compliance in the DBVC Period | Safety | |
| 3.2 Adverso | e Events | | |
| 3.2.1.x | Overall Summary of Treatment-Emergent Adverse Events | Safety | X |
| 3.2.2.x | Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term | Safety | X |
| 3.2.3.x | Summary of Treatment-Emergent Adverse Events by MedDRA Preferred Term in Decreasing Order of Frequency | Safety | X |
| 3.2.4.x | Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class, Preferred Term, and Maximum Severity | Safety | X |
| 3.2.5.x | Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class, Preferred Term, and CTCAE Grade Category | Safety | |
| 3.2.6.x | Summary of Grade 3 or Higher Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term | Safety | X |
| 3.2.7.x | Summary of Grade 3 or Higher Treatment-Emergent Adverse Events by MedDRA Preferred Term in Decreasing Order of Frequency | Safety | X |
| 3.2.8.x | Summary of Serious Treatment-Emergent Adverse Events by MedDRA<br>System Organ Class and Preferred Term | Safety | X |
| 3.2.9.x | Summary of Serious Treatment-Emergent Adverse Events by MedDRA Preferred Term in Decreasing Order of Frequency | Safety | X |
| 3.2.10.x | Summary of Treatment-Related Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term | Safety | X |
| 3.2.11.x | Summary of Treatment-Related Treatment-Emergent Adverse Events by MedDRA Preferred Term in Decreasing Order of Frequency | Safety | X |
| 3.2.12.x | Summary of Grade 3 or Higher Treatment-Related Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term | Safety | |
| 3.2.13.x | Summary of Treatment-Related Serious Treatment-Emergent Adverse<br>Events by MedDRA System Organ Class and Preferred Term | Safety | X |
| 3.2.14.x | Summary of Treatment-Emergent Adverse Events With a Fatal Outcome by MedDRA System Organ Class and Preferred Term | Safety | X |
| 3.2.16.x | Summary of Treatment-Emergent Adverse Events Leading to Dose Interruption by MedDRA System Organ Class and Preferred Term | Safety | X |
| 3.2.17.x | Summary of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug by MedDRA System Organ Class and Preferred Term | Safety | X |
| 3.2.18.x | Summary of Application Site Reactions by MedDRA Preferred Term in Decreasing Order of Frequency | Safety | X |
| 3.3 Labora | tory | | |
| 3.3.1.1.x | Summary of Laboratory Values – Hematology | Safety | X |
| 3.3.1.2.x | Summary of Laboratory Values – Chemistry | Safety | X |
| 3.3.2.1.x | Shift Summary of Hematology Laboratory Values – to the Worst Abnormal Value | Safety | X |
| 3.3.2.2.x | Shift Summary of Chemistry Laboratory Values – to the Worst Abnormal Value | Safety | X |

| Table No. | Title | Population | Standard |
|---|---|---|---|
| 3.3.3.1.x | Shift Summary of Hematology Laboratory Values in CTCAE Grade – to the Worst Grade Abnormal Value | Safety | X |
| 3.3.3.2.x | Shift Summary of Chemistry Laboratory Values in CTCAE Grade – to the Worst Grade Abnormal Value | Safety | X |
| 3.4 Vital Signs | | | |
| 3.4.1.x | Summary of Systolic Blood Pressure | Safety | X |
| 3.4.2.x | Summary of Diastolic Blood Pressure | Safety | X |
| 3.4.3.x | Summary of Pulse | Safety | X |
| 3.4.4.x | Summary of Respiratory Rate | Safety | X |
| 3.4.5.x | Summary of Body Temperature | Safety | X |

Note: For AE tables ending with "x," separate tables will be provided for the DBVC period, OLE period, and the treatment periods (DBVC and OLE periods). For laboratory and vital sign tables ending with "x," separate tables will be provided for the DBVC period and the OLE period.

### **Figures**

| Figure No. | Title | Population |
|---|---|---|
| Efficacy | | |
| 4.1.1.1 | Proportion of Participants Achieving IGA-TS in Treatment Periods | ITT |
| 4.1.1.2 | Proportion of Participants Achieving IGA-TS by Sex in Treatment Periods | ITT |
| 4.1.1.3 | Proportion of Participants Achieving IGA-TS by Baseline Age Group in Treatment Periods | ITT |
| 4.1.1.4 | Proportion of Participants Achieving IGA-TS by Baseline Duration of Disease in Treatment Periods | ITT |
| 4.1.1.5 | Proportion of Participants Achieving IGA-TS by Race in Treatment Periods | ITT |
| 4.1.1.5 | Forest Plot of Response Rate Difference in Achieving IGA-TS at Week 16 | ITT |
| 4.2.1.1 | Proportion of Participants Achieving ITCH4 in Treatment Periods | ITT |
| 4.2.2.1 | Mean and Standard Error Plot of By-Visit Itch NRS Score in Treatment Periods | ITT |
| 4.2.3.1 | Mean and Standard Error Plot of Daily Itch NRS Score from Day 1 to Day 28 | ITT |
| 4.2.4 | Kaplan-Meier Curve of Time to ITCH4 in the DBVC Period | ITT |
| 4.3.1.1 | Mean and Standard Error Plot of By-Visit Skin Pain NRS Score in Treatment Periods | ITT |





# Listings

| Listing No. | Title |
|---|---|
| 2.1 Demogra | 2.1 Demographic and Baseline Characteristics |
| 2.1.1 | Participant Enrollment and Disposition Status |
| 2.1.2 | Participant Inclusion and Exclusion Criteria Violations |
| 2.2 Protocol | 2.2 Protocol Deviations |
| 2.2.1 | Protocol Deviations |
| 2.3 Data Exc | luded From , Efficacy, and/or Safety Analyses |
| 2.3 | Analysis Populations |
| 2.4 Demogra | phic and Baseline Characteristics (Including Prior and Concomitant Medications) |
| 2.4.1 | Demographic and Baseline Characteristics |
| 2.4.2 | Baseline Disease Characteristics |
| 2.4.3 | Medical History |
| 2.4.4 | Prior and Concomitant Medications |
| 2.4.5 | Prior Medications for Cutaneous Lichen Planus |
| 2.5 Drug Exp | posure and Compliance |
| 2.5.1 | Study Drug Exposure and Compliance in the DBVC Period |
| 2.5.2 | Study Drug Exposure in the OLE Period |
| 2.6 Efficacy | |
| 2.6.1 | IGA Score |
| 2.6.2.1 | By-Visit Itch NRS Score |
| 2.6.2.2 | Daily Itch NRS Score |
| 2.6.3.1 | By-Visit Skin Pain NRS Score |
| 2.6.3.2 | Daily Skin Pain NRS Score |
| 2.7 Adverse | Events |
| 2.7.1 | Adverse Events |

| Listing No. | Title |
|---|---|
| 2.7.2 | Adverse Events Leading to Study Drug Discontinuation |
| 2.7.3 | Serious Adverse Events |
| 2.7.4 | Treatment-Related Adverse Events |
| 2.7.5 | Adverse Events With a Fatal Outcome |
| 2.7.6 | Adverse Events Leading to Interruption of Study Drug |
| 2.7.8 | Grade 3 or Higher Adverse Events |
| 2.7.9 | Application Site Reactions |
| 2.8 Laboratory Data | |
| 2.8.1.1 | Clinical Laboratory Values – Hematology |
| 2.8.1.2 | Clinical Laboratory Values – Chemistry |
| 2.8.1.4 | Abnormal Clinical Laboratory Values – Hematology |
| 2.8.1.5 | Abnormal Clinical Laboratory Values – Chemistry |
| Vital Signs | |
| 2.8.2.1 | Vital Signs |
| 2.8.2.2 | Abnormal Vital Sign Values |
| 2.8.2.3 | Alert Vital Sign Values |